CLINICAL TRIAL: NCT04554914
Title: An Open-label, Single-arm, Multicohort, Phase 2 Study to Assess the Efficacy and Safety of Tabelecleucel in Subjects With Epstein Barr Virus Associated Diseases (EBVision)
Brief Title: A Study to Evaluate Tabelecleucel in Participants With Epstein Barr Virus (EBV) Associated Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATA129-EBV-205/F60085DL205; 2024-516623-14-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Epstein-Barr Virus (EBV)-Associated Diseases; EBV+ Lymphoproliferative Disease With Primary Immunodeficiency (EBV+ PID LPD); EBV+ Lymphoproliferative Disease With Acquired (Non-congenital) Immunodeficiency (EBV+ AID LPD); EBV+ Posttransplant Lymphoproliferative Disease in Central Nervous System (EBV+ CNS PTLD); EBV+ Post-transplant Lymphoproliferative Disease (EBV+ PTLD); Solid Organ Transplant Complications; Lymphoproliferative Disorders; Allogeneic Hematopoietic Cell Transplant; Stem Cell Transplant Complications; EBV+ Sarcomas; Leiomyosarcoma
Keywords: Allogeneic, Off-The-Shelf T-cell Immunotherapy; Epstein-Barr Virus (EBV); Epstein-Barr Virus-specific Cytotoxic T lymphocyte (EBV-CTL); Solid Organ Transplant (SOT); Hematopoietic Cell Transplant (HCT); EBVision
MeSH Terms: conditions — Epstein-Barr Virus Infections; Immunologic Deficiency Syndromes; Lymphoproliferative Disorders; Leiomyosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- EBV+ PID LPD (Experimental): Participants with R/R or newly diagnosed EBV+ PID LPD for whom standard first-line therapy is inappropriate, will receive IV tabelecleucel.
  Interventions: Biological: Tabelecleucel
- EBV+ AID LPD (Experimental): Participants with R/R or newly diagnosed EBV+ AID LPD for whom standard first-line therapy is inappropriate, will receive IV tabelecleucel.
  Cohort closed for enrollment after completion of stage1
  Interventions: Biological: Tabelecleucel
- EBV+ CNS PTLD (Experimental): Participants with R/R or newly diagnosed EBV+ CNS PTLD for whom standard first-line therapy is inappropriate, will receive IV tabelecleucel.
  Interventions: Biological: Tabelecleucel
- EBV+ 1L PTLD (inappropriate for first-line therapy or CD20-negative) (Experimental): Participants with EBV+ PTLD for whom standard first-line therapy (rituximab or chemotherapy) is inappropriate, including CD20-negative disease, will receive IV tabelecleucel.
  Interventions: Biological: Tabelecleucel
- EBV+ sarcoma, including LMS, or smooth muscle tumors (Experimental): Participants with newly diagnosed EBV+ sarcoma for whom the standard first-line therapy is inappropriate, including LMS or smooth muscle tumor, will receive IV tabelecleucel.
  Interventions: Biological: Tabelecleucel

INTERVENTIONS:
Biological: Tabelecleucel — Tabelecleucel is being investigated as an off-the-shelf, allogeneic T-cell immunotherapy for the treatment of EBV+ malignancies and diseases.
  Other Names: ATA129; EBV-CTLs

SUMMARY:
The purpose of this study is to assess the efficacy and safety of tabelecleucel in participants with EBV-associated diseases.

DETAILED DESCRIPTION:
This is a multicenter, multicohort, open-label, single-arm, Phase 2 study to assess the efficacy and safety of tabelecleucel for the treatment of EBV-associated diseases. Participants will be enrolled in one of the following cohorts:

* EBV+ lymphoproliferative disease (LPD) in the setting of primary immunodeficiency (PID) (EBV+ PID LPD) that is relapsed and/or refractory (R/R) or newly diagnosed where standard first-line therapy is inappropriate
* EBV+ LPD in the setting of acquired (non-congenital) immunodeficiency (AID) (EBV+ AID LPD) that is R/R or newly diagnosed where standard first-line therapy is inappropriate [cohort closed for enrollment after completion of stage1]
* EBV+ post-transplant lymphoproliferative disease (PTLD) involving the central nervous system (CNS) (EBV+ CNS PTLD) that is R/R or newly diagnosed where standard first-line therapy is inappropriate
* EBV+ PTLD where standard first-line therapy (rituximab or chemotherapy) is inappropriate, including cluster of differentiation antigen 20 (CD20)-negative disease
* EBV+ sarcomas, including leiomyosarcoma (LMS), or smooth muscle tumors that is rapidly progressive where standard first-line therapy is inappropriate

Tabelecleucel will be administered in cycles lasting for 35 days. During each cycle, participants will receive tabelecleucel at a dose of 2 x 10^6 cells/kg intravenously (IV) weekly for 3 weeks, followed by observation through Day 35. Treatment will continue until maximal response, disease progression, unacceptable toxicity, or initiation of nonprotocol therapy for the underlying disease. For EBV+ sarcoma cohort, treatment will continue until disease progression, unacceptable toxicity, two consecutive complete responses (CRs), or up to 12 months from the first dose. Participants who fail to respond to initial tabelecleucel treatment may continue tabelecleucel with a different human leukocyte antigen (HLA) restriction (termed a Restriction Switch), if available; administration of tabelecleucel with up to four different HLA restrictions is allowed for any participant.

After treatment is completed or discontinued, participants will complete a safety follow-up visit at 30 days after the last dose and then will enter a quarterly follow-up period. Participants without documented disease progression will be assessed every 3 months after the safety follow-up visit for continued evaluation of disease response until the end of study (EOS) visit at which occurs at 12 (± 1) months after Cycle 1 Day 1 for adults, and 24 (± 1) months after Cycle 1 Day 1 for pediatric participants. Participants with disease progression any time prior to the EOS visit will continue to be followed every 3 months for survival status until the EOS visit.

An adaptive 2-stage design will be used for each relevant cohort in this study. For each cohort, 8 evaluable participants will be enrolled in Stage 1. The decision to move to Stage 2 enrollment will be based on an interim analysis of the first 8 evaluable participants in the cohort using investigator's assessment (per defined radiologic, clinical, and/or laboratory response criteria) who receive tabelecleucel and have at least 1 valid postbaseline disease response assessment. The number of participants enrolled in Stage 2 for each cohort will depend on the number of observed responders in Stage 1. Sponsor may decide not to move forward to Stage 2 in any cohort even if the criteria to move forward for that cohort are met. The decision not to move forward may also be based on data from one or other cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of EBV+ disease.
* Eastern Cooperative Oncology Group performance status ≤ 3 for participants aged ≥ 16 years; Lansky score ≥ 20 for participants from ≥ 1 year to < 16 years.
* Adequate organ function test results, unless organ dysfunction is considered to be due to the underlying EBV-associated disease by the investigator.

Cohort-specific Inclusion Criteria:

* For participants with CNS PTLD:

  * R/R or newly diagnosed EBV+ CNS PTLD for whom the standard. first-line therapy is inappropriate, as determined by the investigator. The CNS PTLD is histologically confirmed by at least biopsy-proven EBV+ CNS PTLD or positive CSF cytology with or without radiographically measurable intracranial disease with EBV detected in CSF.
  * Participants with R/R disease must have had at least one prior line of systemic therapy and one of the following: radiographic disease progression per Lugano Classification during or after treatment or failure to achieve a CR or PR (defined by Lugano radiographic criteria) after standard first-line therapy.
  * Participant may have systemic and CNS disease or CNS disease only.

Exclusion Criteria:

* Currently active Burkitt, T-cell, natural killer/T-cell lymphoma/LPD, Hodgkin, plasmablastic, transformed lymphoma, active hemophagocytic lymphohistiocytosis, or other malignancies requiring systemic therapy.
* Serious known active infections, defined as ongoing uncontrolled adenovirus infection or infections requiring systemic therapy at the time of enrollment, or known history of human immunodeficiency virus (HIV) infection.
* Suspected or confirmed Grade ≥ 2 acute graft-versus-host disease (GvHD) per the Center for International Blood and Marrow Transplant Research (CIBMTR) consensus grading system or extensive chronic GvHD per National Institutes of Health (NIH) consensus criteria at the time of the enrollment.
* Need for vasopressor or ventilatory support at the time of enrollment.
* Prior therapy (in order of increasing washout period) prior to enrollment as follows:

  * Within 4 weeks or 5 half-lives (whichever is shorter) for any investigational product and/ or any chemotherapy (systemic or intrathecal), targeted small molecule therapy, or antibody/biologic therapy. Note: prior anti-CD20 antibody use is permitted within the washout period if a subsequent disease response assessment indicates disease progression.
  * Within 8 weeks: prior tabelecleucel (> 8 weeks prior to enrollment) is permitted if response was obtained or if usual protocol-directed therapeutic options were not exhausted, for cellular therapies (chimeric antigen receptor therapies directed at T-cells or T-cell subsets, donor lymphocyte infusion, other CTLs or virus-specific T-cells); and/or therapies which could impact tabelecleucel function (anti-thymocyte globulin, alemtuzumab).
  * Any prior treatment with EBV-CTLs with the exception of tabelecleucel as above
* Women who are breastfeeding or pregnant.
* Unwilling to comply with protocol specified contraceptive/reproductive restrictions from enrollment through 90 days after the last treatment.
* Inability or unwillingness to comply with all study procedures.
* Ongoing need for daily steroids of > 0.5 mg/kg prednisone or glucocorticoid equivalent, ongoing methotrexate, or extracorporeal photopheresis (for participants with CNS disease, protocol-specified dexamethasone is permitted and concludes by the time of enrollment).
* Any conditions that may put the study outcomes at undue risk (life expectancy < 60 days or any life-threatening illness, medical condition, or organ system dysfunction).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
Duration of response (DOR) | Up to 2 years
Progression-free survival (PFS) | Up to 2 years
For EBV+ PID LPD cohort: Number of participants who reach definitive therapy (ie, allogeneic HCT) for the underlying disease | Up to 2 years
For EBV+ PID LPD cohort: Time to definitive therapy | Up to 2 years
For EBV+ sarcoma cohort, including LMS, or smooth muscle tumors: Clinical benefit rate | Up to 2 years
For EBV+ sarcoma cohort, including LMS, or smooth muscle tumors: ORR by immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria | Up to 2 years
Number of Participants who Experience Adverse Events (AE) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anke Friedetzky, Study Director — Pierre Fabre Laboratories
Locations (40):
- United States (23):
  - University of California Los Angeles (UCLA) (Adults and Pediatrics), Los Angeles, California
  - Children's Hospital of Orange County (Pediatrics [up to 25 years old]), Orange, California
  - Lucile Packard Children's Hospital Stanford (Pediatrics only), Palo Alto, California
  - University of California Davis Comprehensive Cancer Center (Adults and Pediatrics), Sacramento, California
  - Sylvester Comprehensive Cancer Center/ University of Miami, Miami, Florida
  - Moffit Cancer Center (Adults only), Tampa, Florida
  - Children's Healthcare of Atlanta (Pediatrics only [up to 25 years old]), Atlanta, Georgia
  - Emory University/Winship Cancer Institute (Adults [>= 16 years]), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago (Pediatrics only), Chicago, Illinois
  - University of Maryland Medical Center (Adults only), Baltimore, Maryland
  - Dana Farber Cancer Institute (DFCI) (Adults and Pediatrics), Boston, Massachusetts
  - University of Michigan Rogel Cancer Center (Adults and Pediatrics), Ann Arbor, Michigan
  - University of Minnesota (Adults only), Minneapolis, Minnesota
  - Washington University in St. Louis (Adults only), St Louis, Missouri
  - Columbia University Irving Medical Center (Adults only), New York, New York
  - Memorial Sloan-Kettering Cancer Center (Adults and Pediatrics), New York, New York
  - The Children's Hospital at Montefiore (Adults and Pediatrics), The Bronx, New York
  - Cleveland Clinic Taussig Cancer Center (Adults and Pediatrics), Cleveland, Ohio
  - The Ohio State University - The James Cancer Hospital and Solove Research Institute (Adults only), Columbus, Ohio
  - Oregon Health and Science University (Adults and Pediatrics), Portland, Oregon
  - Medical University of South Carolina (Adults and Pediatrics), Charleston, South Carolina
  - University of Texas Southwestern Medical Center (Pediatrics only), Dallas, Texas
  - MD Anderson (Adults and Pediatrics), Houston, Texas
- Austria (3):
  - Uniklinikum Salzburg Landeskrankenhaus (Adults only), Salzburg, Salzburg
  - Medizinische Universität Graz (Adults only), Graz, Styria
  - Medizinische Universität Wien (Adults only), Vienna, Vienna
- Belgium (3):
  - Hôpital Universitaire des Enfants Reine Fabiola (Pediatrics only), Brussels, Brussles
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan (Adults only), Bruges, West-Vlaanderen
  - Algemeen Ziekenhuis Delta - Campus Rumbeke (Adults only), Roeselare, West-Vlaanderen
- France (3):
  - Hôpital Saint-Eloi (Adults and Pediatrics), Montpellier, Montpellier
  - Hôpital Necker-Enfants Malades (Adults and Pediatrics), Paris, Paris
  - Hôpital Universitaire Pitié Salpêtrière (Adults only), Paris
- Italy (3):
  - Azienda Ospedaliero-Universitaria Pisana (Adults only), Pisa, Pisa
  - Ospedale Pediatrico Bambino Gesù (Adults and Pediatrics), Roma, Roma
  - Ospedale Infantile Regina Margherita (Pediatrics only), Torino, Torino
- Spain (3):
  - Hospital Universitari Vall d'Hebrón (Adults and Pediatrics), Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal (Adults only), Madrid, Madrid
  - Hospital Universitario Virgen del Rocio (Adults and Pediatrics), Seville, Sevilla
- United Kingdom (2):
  - University Hospital Birmingham NHS Foundation Trust (Adults only), Birmingham, England
  - Great Ormond Street Hospital (Pediatrics only), London, England

IPD SHARING:
Plan to Share IPD: No